CLINICAL TRIAL: NCT03581045
Title: Postural Control Under Different Cognitive Loads in Adult Survivors of Acute Lymphoblastic Leukemia and Age-Matched Healthy Individuals
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PCALL; NCI-2018-01471 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2018-06-18; First posted 2018-07-10 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; ALL; Survivors; Cognitive performance; Postural control
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALL Survivors: Adult survivors of Acute Lymphoblastic Leukemia (ALL) enrolled on the SJLIFE protocol
- Control Group: Healthy Individuals with no history of childhood or adult onset cancer, matched on age- and sex

SUMMARY:
The purpose of this study is to determine if adult survivors of childhood Acute Lymphoblastic Leukemia (ALL) enrolled on the SJLife (St. Jude Life) protocol are at increased risk for postural control deficits compared to individuals with no cancer history. All participants will be assessed for their ability to maintain an upright posture, walk at their usual speed, and to tandem walk, all while engaged in a cognitive task.

Primary Objective

To compare changes in postural control in ALL survivors to changes in postural control in healthy controls, matched on age- and sex- in simple versus complex standing and walking activities (complex: standing or walking with added cognitive load).

Secondary Objective

To identify demographic and performance related risk factors for decreased postural control during complex standing or walking activities in survivors and controls and to evaluate associations between treatment and the changes in postural control during complex activities among survivors.

DETAILED DESCRIPTION:
Cognitive performance (attention and working memory) will be evaluated using the auditory N-Back test. The 0-back condition and the 2-back condition will be used. After cognitive assessment, participants will perform 3 different postural control tasks (standing balance, regular gait, and tandem gait) in a random order. Postural tasks for each participant will be determined by using random allocation envelopes.

Computerized dynamic posturography will be used to evaluate standing balance with no added cognitive load. Standing balance assessment will be repeated two more times, once with participants engaged in performing the auditory 0-back task, and then with simultaneously performing the auditory 2-back task. Regular gait at participants' preferred speed will be examined using 6 light-weight wearable inertial sensors. The regular walking assessment will be repeated with simultaneous performance of the 0-back task and then with simultaneous engagement in the 2-back task. We have also included a tandem gait (placing one foot directly in front of the other) in order to make the postural task more challenging. The wearable inertial sensors will be used to record participants' gait characteristics while tandem walking. The tandem walk assessment will be repeated once with the participant simultaneously perform the 0-back task and then with the 2-back task. The estimated required time to perform all of the assessments and with inclusion of 3 rest intervals is 2 hours.

In addition, data from the overall SJLIFE assessment will be used in analysis.

ELIGIBILITY:
Inclusion Criteria - Cases:

* Diagnosis of childhood ALL
* At least 5 years post ALL diagnosis
* No history of secondary malignancies after an ALL diagnosis
* Enrollment on the SJLIFE protocol
* Ages 18.00 to 39.99
* Ability to stand and walk for 20 seconds or more
* Ability to answer the eligibility questions
* Ability to provide informed consent

Inclusion Criteria - Controls:

* No history of childhood or adult onset cancer
* Enrollment on the SJLIFE protocol
* Ages 18.00 to 39.99
* Ability to stand and walk for 20 seconds or more
* Ability to answer the eligibility questions
* Ability to provide informed consent

Inclusion of Women and Minorities:

• Male and females of all races and ethnic groups are eligible

Exclusion Criteria:

* Currently receiving treatment for cancer
* Weight ≥ 300 lb (the balance system has a weight limit)
* Does not speak English
* Self-reports of hearing issues
* Pregnant females
* Inability or unwillingness of research participant to give written informed consent.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population will include 50 Adults survivors of childhood Acute Lymphoblastic Leukemia (ALL) enrolled on the SJLife protocol, and 50 healthy controls matched on age- and sex.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Regular gait speed | Up to 1 hour
  Regular gait will be evaluated in three different testing conditions: regular gait assessment while participants are engaged in performing a challenging cognitive task (2-back), regular gait assessment while participants are engaged in performing an easy cognitive task (0-bak) and regular gait assessment with no additional cognitive load (baseline). In each condition, the difference in gait speed of each survivor and his/her matched control will be obtained. Then the obtained differences at regular gait assessment with no additional cognitive load (baseline) and regular gait while performing the challenging cognitive task (2-bck) will be compared using a paired t-test.
Composite score from standing balance test | Up to 1 hour
  Standing balance ability will be examined in three different testing conditions: standing balance while participants are engaged in performing a challenging cognitive task (2-back), standing balance while participants are engaged in performing an easy cognitive task (0-back), and standing balance assessment with no additional cognitive load. In each condition, the difference in composite score of each survivor and his/her matched control will be obtained. Then the obtained differences at standing balance assessment with no additional cognitive load (baseline) and standing balance assessment while performing the challenging cognitive task (2-back) will be compared using a paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Ness, PhD, Principal Investigator — St. Jude Children's Reearch Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols